CLINICAL TRIAL: NCT04572282
Title: Single Arm Pilot Study on a Mobile App for Symptoms Monitoring in Cancer Patients on Active Treatments
Brief Title: Mobile App for Symptoms Monitoring in Cancer Patients: a Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Associacao de Investigacao de Cuidados de Suporte em Oncologia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 3
Record Dates: First submitted 2020-09-12; First posted 2020-10-01 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-09

CONDITIONS: Cancer; Symptoms and Signs; Quality of Life; Chemotherapeutic Agent Toxicity
Keywords: cancer; quality of life; digital healthcare; remote monitoring; symptoms; supportive care; cancer survivors
MeSH Terms: conditions — Neoplasms; Signs and Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mentora (Experimental): Remote symptoms monitoring with mobile app
  Interventions: Device: Mentora app

INTERVENTIONS:
Device: Mentora app — Remote monitoring mobile app

SUMMARY:
With the growing number of cancer survivors, challenges to deal with comorbidities and impacted quality of life of cancer survivors by the disease and treatments also surge. Symptoms and Adverse Events are common and insufficiently monitored in real time / real life, which leads to increased symptom burden, treatment delays and unplanned hospital admissions. Remote monitoring apps have been shown to improve quality of life, symptom control and survival in published clinical trials, but no data with such interventions exists on the Portuguese population.

We will conduct a pilot study to explore the feasibility of a mobile app for remote symptom monitoring in cancer patients. Patients will be recruited in Portuguese hospitals and will be invited to test the app for one month. Patient experience and satisfaction will be assessed via a weekly survey.

The results of this pilot study will inform subsequent randomized clinical trials to test safety and efficacy of remote monitoring and lifestyle interventions to improve symptoms control and quality of life.

DETAILED DESCRIPTION:
This is a single cohort study on cancer patients to explore the feasibility of mobile app for symptom monitoring and inform future randomized clinical trials and implementation. Patients will be screened at oncology visits for inclusion criteria and will be invited to use a mobile app to monitor and track treatment side-effects.

We will recruit a minimum of 10 cancer patients under systemic anti-neoplasic treatment being followed in medical oncology departments in portuguese hospitals. between February 1st and March 30th.

Participants will be invited to register their treatment side effects and symptoms on a health app designed for this purpose.

The Mentora Health App include a PRO-CTCAE™ based tool (a patient-reported outcome measurement system developed by the National Cancer Institute), version 1.1, that includes 80 symptoms (attachment 1) and has been translated and validated to Portuguese (Portugal) by the authoring entity. These symptoms are graded on a five-point scale from 0 (not present) to 4 (disabling) based on clinical criteria.

ELIGIBILITY:
Inclusion Criteria:

* adults (18 years old or older)
* with a cancer diagnosis at any stage of any primary tumor (solid or hematologic)
* in systemic oncologic treatments of any type (including but not limited to immunotherapy, chemotherapy and targeted therapies) expected to continue for at least 4 weeks after enrolment, except when single treatment with hormone therapy for prostate cancer or breast cancer
* fluent in written Portuguese
* with a personal mobile smartphone (android or iphone)
* willing to give informed consent for study participation

Exclusion criteria:

* Cognitive impairment or disability that limits capacity to comply with study interventions and assessments as per attending physician's evaluation
* Having a life expectancy < 3 months as determined by the attending oncologist ECOG performance status greater than 2
* Unable to read and comprehend written portuguese language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Compliance rates with the weekly reports or weekly symptom log on the app higher than 60%% (Acceptability of the MHapp) | 1 month
  acceptability of the MHapp, measured by adherence to self-reporting will be assessed at 1 month. The outcome will be considered positive if at least one of the 2 following criteria applies to more than 60% of participants enrolled: replies to 2 or more weekly reports OR at least one weekly log to the app.

SECONDARY OUTCOMES:
% of side effects and adverse events reported on medical appointments also registered in the MHapp | 1 month
  % of side effects and adverse events reported on medical appointments also registered in mh
Total attendance - retention rate/total withdraw from study (30 days) | 1 month
  Total attendance - retention rate/total withdraw from study (30 days)
Impact of MHapp on cancer QoL (EORTC quality of life c 30): comparison between baseline, and 1 month | 1 month
  Higher values after the 1 month intervention mean positive impact with increased quality of life
Report healthcare resources use: number of unplanned hospital visits or calls; unplanned hospitalizations; time inside medical appointments | 1 month
  number of unplanned hospital visits or calls; unplanned hospitalizations; time inside medical appointments
Frequency of grade 3 and 4 adverse events | 1 month
  Number of grade 3 and 4 adverse events reported
Satisfaction of clinical oncology doctors and nurses with the information report provided by the MHapp on a Likert scale from 0 (not satisfied at all) to 7 (Very satisfied) and through qualitative analysis of open ended questions | 1 month
  Satisfaction of clinical oncology doctors and nurses with the information report provided by the MHapp on a Likert scale from 0 (not satisfied at all) to 7 (Very satisfied) and through qualitative analysis of open ended questions

CONTACTS AND LOCATIONS:
Overall Officials: Catarina Ribeiro, Principal Investigator — Associacao de Investigacao de Cuidados de Suporte em Oncologia

IPD SHARING:
Plan to Share IPD: No